CLINICAL TRIAL: NCT05109754
Title: Home Non-Invasive Ventilation Targeting Expiratory Flow Limitation in Severe Hypercapnic COPD.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Devices not available
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Marta Kaminska, Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022-8261
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPAP EFL (Experimental): Phase 1: use device for 2 months
  Phase 2: use device for 12 months
  Interventions: Device: BiPAP EFL

INTERVENTIONS:
Device: BiPAP EFL — Non-invasive ventilation using a novel ventilatory mode targeting expiratory flow limitation in COPD

SUMMARY:
In this 2-phase pilot study, the BiPAP A40 EFL will be evaluated in patients with severe COPD requiring home non-invasive ventilatory support with respect to patient-related and physiologic outcomes.

DETAILED DESCRIPTION:
Objective phase 1: in patients with COPD already established on home NIV, to assess the effect of 2 months of the A40EFL on ventilator parameters, physiologic and patient-related outcomes (PRO), in comparison to the patients' usual settings as prescribed by their treating physician.

The two primary outcomes will be the nightly duration of NIV use and NIV-related symptoms (S3-NIV questionnaire). Patient preference will be a secondary outcome.

Objective phase 2 : In hypercapnic patients with COPD with a prior hypercapnic exacerbation requiring NIV in hospital, to obtain preliminary data regarding the impact of home NIV using the A40EFL on COPD exacerbations and physiologic and patient-related outcomes.

The primary outcome will be the number of hospitalizations over 12 months on A40EFL.

Secondary outcomes will include descriptive data on number of exacerbations not requiring hospitalization but treated with antibiotics or prednisone.

Additional secondary outcomes, physiologic and PRO, for both phases 1 & 2, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1:

severe COPD with FEV1<50%, using home NIV successfully for at least 2 months through the Quebec National Program for Home Ventilatory Assistance (NPHVA).

* Phase 2:

severe COPD with FEV1<50%; pCO2>= 52 on arterial or capillary blood gas measured 2-4 weeks after acute NIV use and discontinuation

Exclusion Criteria:

* Phase 1

COPD exacerbation requiring treatment (including hospitalization) within the last 6 weeks; surgical procedure or major illness within the last 3 months; kyphoscoliosis, neuromuscular disease, other lung disease (e.g. fibrosis); active cancer; expected survival < 2 months; listed on the transplant list.

* Phase 2:

any additional condition potentially predisposing to hypercapnia such as: obesity (BMI> 30kg/m2), kyphoscoliosis, neuromuscular disease, other lung disease (e.g. fibrosis), severe obstructive sleep apnea (AHI>30/h on prior testing if available, but will not test as part of the study); active cancer; expected survival < 2 months; listed on the transplant list at start of study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The nightly duration of Non-Invasive Ventilation use | 2 months
  (Phase 1)
  Measured in hours and minutes.
S3-NIV (Non-Invasive Ventilation) questionnaire score | 2 months
  NIV-related symptoms (Phase 1) Dupuis-Lozeron E, Gex G, Pasquina P, et al. Development and validation of a simple tool for the assessment of home noninvasive ventilation: the S3-NIV questionnaire. Eur Respir J 2018; 52: 1801182.
  The lowest score corresponds to highest adverse impact of disease and treatment.
The number of hospitalizations during the study period, compared with year prior to inclusion | 12 months
  (phase 2)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Kaminska, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- MUHC, Montreal, Quebec, Canada